CLINICAL TRIAL: NCT06072924
Title: Impact of Lingual Endurance Exercise on Rehabilitation of Swallowing Impairments After Ischemic Stroke
Brief Title: K01 Impacts of Lingual Endurance Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); TriHealth Inc. (Other)
Responsible Party: Principal Investigator, Brittany Krekeler, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0582 Lingual Endurance; 1K01HD111680-01 (NIH)
Record Dates: First submitted 2023-09-19; First posted 2023-10-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Dysphagia; Dysphagia, Oropharyngeal; Ischemic Stroke; Stroke
Keywords: swallowing trouble; difficulty swallowing; swallow rehab
MeSH Terms: conditions — Deglutition Disorders; Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Randomized Sham Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lingual Endurance Exercise (Experimental): The experimental exercise group will participate in 3 training sessions per day for 8 weeks. Endurance exercise will include completing isotonic endurance repetitions 3 times a day. Number of repetitions per session will be determined during baseline testing, and re-evaluated every 2 weeks, for each participant.
  Interventions: Behavioral: Isotonic Endurance Exercise
- Sham Exercise (Sham Comparator): The sham control group will be instructed to press the lingual sensor 30 times at a very low-pressure threshold (approximately 1-15 kPa), which will be monitored weekly via device output sent to the study team to avoid use of excessive force that would qualify as exercise.
  Interventions: Behavioral: Sham Exercise

INTERVENTIONS:
Behavioral: Isotonic Endurance Exercise — Pressing tongue against a pressure sensor at the set number of repetitions per session (individualized per participant) 3 times per day
  Arms: Lingual Endurance Exercise
Behavioral: Sham Exercise — Pressing tongue against pressure sensor at a low threshold (1-15kPa) 30x/day
  Other Names: Learning group
  Arms: Sham Exercise

SUMMARY:
The goal of this clinical trial is to learn whether a tongue endurance exercise program can improve swallowing function in adults with dysphagia after a stroke. It also aims to explore how this exercise may affect brain structure and connectivity involved in swallowing. The main questions it aims to answer are:

Primary Aim: Does lingual endurance exercise improve swallowing function compared to a sham therapy? Secondary Aim: Does lingual endurance exercise lead to changes in brain structure or neuroplasticity, as measured by MRI?

Researchers will compare a group receiving tongue endurance exercises to a sham therapy group to see whether the treatment improves tongue function, swallowing.

Participants will:

* Complete a baseline swallowing assessment and MRI
* Be randomly assigned to either the lingual exercise or sham therapy group
* Complete 8 weeks of home-based tongue exercise therapy
* Return for follow-up swallowing assessments
* A subgroup of participants will complete a pre-treatment and post-treatment MRI.

DETAILED DESCRIPTION:
This randomized, controlled clinical trial investigates the efficacy of a 8-week lingual endurance exercise program in adults with dysphagia following stroke. The study uses a two-arm, parallel-group design with participants randomized to either a lingual endurance exercise group or a sham therapy control group. Both interventions are delivered using a lingual manometer, which participants use at home under monitored conditions.

The primary aim is to evaluate changes in oral-phase swallowing physiology using the Modified Barium Swallow Impairment Profile (MBSImP) Oral Total Score, as assessed through video-fluoroscopic swallowing study (VFSS).

An exploratory aim will assess potential neuroplasticity associated with lingual endurance exercise using multimodal neuroimaging. Participants who meet MRI eligibility criteria undergo pre- and post-intervention imaging, including diffusion tensor imaging (DTI) to assess white matter integrity, high-resolution structural imaging for cortical thickness estimation, and functional MRI (task-based and resting state). Data will be used to evaluate intervention-related changes in regions associated with swallowing motor control and sensory integration.

This study also supports the investigator's training in clinical trial methodology, swallowing outcomes analysis, and neuroimaging techniques, and will inform a future, fully powered efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* 1) 3-6 months since most recent diagnosis of ischemic, confirmed from clinical imaging) with or without small hemorrhagic transformation (HI-1)
* 2) Have some indication of on-going swallowing issues
* 3) English Speaking

Exclusion Criteria:

* 1) ≤18 years of age
* 2) history of dysphagia prior to or after the stroke caused by any of the following conditions: gastrointestinal disease, traumatic brain injury, head and neck cancer, surgery involving the pharynx or larynx
* 3) history of other neurological disease (i.e. multiple sclerosis, ALS, Parkinson's, dementia).
* 4) Medium to large hemorrhagic transformation/involvement documented on clinical stroke imaging 5) 5) History of temporomandibular joint and muscle disorders (also known as TMJ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Modified Barium Swallow Study Impairment Profile Oral Total (MBSImP OT Score) | Change from Baseline (at the end of 8 weeks)
  MBSImP is a validated, standardized tool for assessing oral, pharyngeal, and esophageal swallowing function. We will be using change in OT score (sum of components 1-6) as our primary outcome measure.

SECONDARY OUTCOMES:
Pharyngeal Swallow Efficiency | Change from Baseline (at the end of 8 weeks)
  Measurements via the ASPEKT method (Analysis of Swallowing Physiology: Events, Kinematics, and Timing) will be analyzed to compared pre and post treatment swallow efficiency. The amount will be presented as a percent of anatomical C2-C4 Scalar. Higher percentile, in general indicated greater impairment, however these will be compared to published normative data for reference.
Penetration Aspiration Scale (PAS) Scores | Change from Baseline (at the end of 8 weeks)
  8-point rating scale that is used to capture both degree and sensation of penetration and aspiration.
Adherence | At the end of 8 weeks
  number of repetitions attempted/total number of repetitions prescribed
Pharyngeal Swallow Safety | Change from Baseline (at the end of 8 weeks)
  Closure above the airway must be achieved for swallowing safety and in a timely manner. The ASPEKT method (Analysis of Swallow Physiology: Events, Kinematics and Timing) will be used to analyze changes of laryngeal vestibule closure pre and post treatment.
Maximum Isometric Pressure imaging with video-fluoroscopy | Change from Baseline (at the end of 8 weeks)
  Maximum isometric press will be recorded in kPa and with recorded imaging using video-fluoroscopy. This will be collected pre- and post-therapy to determine any changes in oropharyngeal movements with a lingual press.
Dietary Intake (Average Daily Calorie Intake) Outcome | Change from Baseline (at the end of 8 weeks)
  A pre treatment and post treatment 24 hour dietary recall will be collected in a subset or participants. This information will be used for estimating nutrient and food group intake to characterize usual diet and to assess changes over time. Nutrition Data Systems for Research (NDSR) (Nutrition Coordinating Center, University of Minnesota, Minneapolis, MN) software and foods database will be used to assess average daily energy (kJ) intake over 3 days
Food Textures Consumed Outcome | Change from Baseline (at the end of 8 weeks)
  A pre treatment and post treatment 24 hour dietary recall will be collected in a subset or participants. This information will be used for estimating nutrient and food group intake to characterize usual diet and to assess changes over time. Nutrition Data Systems for Research (NDSR) (Nutrition Coordinating Center, University of Minnesota, Minneapolis, MN) software and foods database will be used to assess the relative percentage (%) of dry texture food intake, on average, across three days

OTHER OUTCOMES:
Change in fractional anisotropy (FA) | Change from Baseline (at the end of 8 weeks)
  Diffusion Tensor Imaging (DTI) has been the most common analysis framework that is used to analyze the signal from diffusion MRI (dMRI) to gather information about the properties of the underlying white matter.
Change in cortical thickness | Change from Baseline (at the end of 8 weeks)
  Diffusion Tensor Imaging (DTI) has been the most common analysis framework that is used to analyze the signal from diffusion MRI (dMRI) to gather information about the properties of the underlying white matter.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany N Krekeler, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan currently to share IPD with other researchers.